CLINICAL TRIAL: NCT00231426
Title: Arrhythmia Single Shock DFT Versus ULV: Risk Reduction Evaluation With ICDs Study
Brief Title: ASSURE Study - Arrhythmia Single Shock DFT Versus ULV: Risk Reduction Evaluation With ICD Implantations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR-CA-031203-M
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Tachyarrhythmia
MeSH Terms: conditions — Tachycardia

INTERVENTIONS:
Device: ICD

SUMMARY:
The ASSURE Study will evaluate shock conversion performance when programming the first shock of an implantable cardioverter-defibrillation (ICD) is based on an implant test consisting of either 1) a single induction of ventricular fibrillation (VF) and subsequent demonstration conversion success at 14 J or 2) an upper limit of vulnerability (ULV) test at 14 J.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for an ICD including cardiac resynchronization therapy (CRT) devices
* Patients who sign and date a Patient Informed Consent form prior to the implant visit
* Patients who remain in the clinical care of the enrolling physician in approved centers
* Patients who receive only left-sided pectoral implantations with the ICD lead placed in the right ventricular apex
* Patients who have a minimum R wave of at least 7 mV; or for ICD replacement, patients who have a minimum chronic R wave of at least 5 mV

Exclusion Criteria:

* Patients who are involved in Non-Invasive Programming Stimulation (NIPS) studies
* Patients who undergo lead repositioning
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients who have or who are likely to receive a tricuspid valve prosthesis
* Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study
* Patients who are younger than 18 years of age
* Patients who are pregnant or plan to become pregnant during the study
* Patients whose life expectancy is less than 12 months
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: John D Day, M.D., Principal Investigator — LDS Hospital, Salt Lake City, Utah
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States